CLINICAL TRIAL: NCT04219891
Title: Pivotal Trial of WaveLight® EX500 Excimer Laser System for the Correction of Myopia With and Without Astigmatism Using InnovEyes™ in Conjunction With InnovEyes™ Sightmap
Brief Title: WaveLight® EX500 Excimer Laser System for the Correction of Myopia Using InnovEyes™ in Conjunction With InnovEyes™ Sightmap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFP911-C001
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Myopia
Keywords: LASIK; Ray Tracing; Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- WaveLight EX500 excimer laser system (Experimental): Laser-assisted in situ keratomileusis (LASIK) surgery using the WaveLight EX500 excimer laser with InnovEyes software in conjunction with InnovEyes sightmap
  Interventions: Device: WaveLight EX500 excimer laser system with InnovEyes sightmap; Procedure: LASIK; Device: InnovEyes sightmap

INTERVENTIONS:
Device: WaveLight EX500 excimer laser system with InnovEyes sightmap — FDA approved stationary scanning-spot excimer laser system used during refractive surgery for the treatment of myopia, myopic astigmatism, hyperopia, hyperopic astigmatism, and mixed astigmatism. For this clinical study, the WaveLight EX500 software will be upgraded to include the InnovEyes treatment.
Procedure: LASIK — Procedure that reshapes the front part of the eye (cornea) so that light traveling through it is properly focused on the back part of the eye (retina). The procedure will be performed using the WaveLight EX500 excimer laser system and data obtained from the InnovEyes sightmap.
Device: InnovEyes sightmap — Non-contact ophthalmic diagnostic device that captures images of the eye and collects ocular data preoperatively to generate a patient-specific ablation profile for refractive correction surgery

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the WaveLight EX500 excimer laser system for the correction of myopia with and without astigmatism using InnovEyes in conjunction with InnovEyes sightmap.

DETAILED DESCRIPTION:
Qualified subjects will receive treatment in both eyes and be followed for 1 year. Subjects will be asked to attend a total of 9 visits (Screening, Day 0 Surgery, Day 1, Week 1, Month 1, Month 3, Month 6, Month 9, and Year 1). The primary endpoints will be assessed at refractive stability, defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at 3 months after surgery when compared with the 1-month visit) that meets all the protocol-specified stability requirements. Total expected duration of subject participation is approximately 1 year. This study will be conducted in the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Myopia up to and including -11.00 D with or without astigmatism up to -4.50 D, with MRSE no more than -12.00 D
* Best corrected photopic distance visual acuity of 20/20 or better
* Uncorrected photopic distance visual acuity of 20/40 or worse
* Stable refraction (within ± 0.50 D) as determined by MRSE for a minimum of 12 months prior to surgery

Key Exclusion Criteria:

* History or evidence of active or inactive corneal disease or retinal vascular disease, keratoconus or glaucoma (or suspect)
* Previous intraocular or corneal surgery
* Intent to have monovision treatment

Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Surgical, Study Director — Alcon Research
Locations (9):
- United States (9):
  - Alcon Investigative Site, San Diego, California
  - Price Vision Group, Indianapolis, Indiana
  - Alcon Investigative Site, Chevy Chase, Maryland
  - Alcon Investigative Site, Kansas City, Missouri
  - Alcon Investigative Site, St Louis, Missouri
  - Alcon Investigative Site, Omaha, Nebraska
  - Alcon Investigative Site, Mt. Pleasant, South Carolina
  - Alcon Investigative Site, Sioux Falls, South Dakota
  - Alcon Investigative Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 9 investigative sites located in 1 country (US).
Pre-assignment Details: Of the 272 enrolled, 104 participants were exited prior to treatment as screen failures. This reporting group includes all subjects with attempted surgery (168 subjects / 336 eyes).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | WaveLight EX500 Excimer Laser System
Started (Attempted Surgery) | 168; 336 eyes
Successful Surgery | 168; 336 eyes
Safety Analysis Set (SAS) (All eyes that undergo surgery or attempted surgery (defined as eye drops given for flap treatment)) | 168; 336 eyes
Full Analysis Set (FAS) (All eyes that successfully undergo surgery, with one subject excluded due to pregnancy) | 167; 334 eyes
FAS at Refractive Stability (Refractive Stability was considered to be achieved at the Month 3 visit.) | 163; 236 eyes
Completed | 163; 326 eyes
Not Completed | 5; 10 eyes
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 167
Number analyzed (eyes) | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 128
  Black or African American | 10
  American Indian or Alaska Native | 1
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 1
  Multi-Racial | 2
  Other | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 143
  Not reported | 1
  Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) of 20/40 or Better (in Eyes With Preoperative Best Corrected Distance Visual Acuity (BCDVA) of 20/20 or Better) at Refractive Stability
Description: Visual acuity (VA) was assessed using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts at a distance of 4 meters and reported in Snellen, where 20/20 indicates normal distance eyesight. Preoperatively, VA was assessed with correction in place. Postoperatively, VA was assessed with no correction in place. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive stability was considered to be achieved at the Month 3 visit. A higher percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Preoperative Visit (Day -30 to Day -1), Month 1, Month 3
Population: FAS. Note: 1 eye was excluded from this analysis due to not having a preoperative best corrected distance visual acuity (BCDVA) of 20/20 or better.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 163
Number analyzed (eyes) | 325
percentage of eyes | 100.0

2. Primary Outcome: Percentage of Eyes With Manifest Refractive Spherical Equivalent (MRSE) Within +/- 0.50 Diopter (D) at Refractive Stability
Description: A manifest refraction (manual refraction) was performed using a phoropter. The spherical equivalent was calculated by adding the sum of the sphere power with half of the cylinder power and reported in diopters. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive Stability was considered to be achieved at the Month 3 visit. A higher percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Month 1, Month 3
Population: FAS
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 163
Number analyzed (eyes) | 326
percentage of eyes | 92.0

3. Primary Outcome: Percentage of Eyes With MRSE Within +/- 1.00 D at Refractive Stability
Description: as for outcome 2
Time Frame: Month 1, Month 3
Population: FAS
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 163
Number analyzed (eyes) | 326
percentage of eyes | 98.5

4. Primary Outcome: Percentage of Eyes That Achieve Refractive Stability Assessed as Change From Baseline in MRSE of Equal to or Less Than 1.0 D
Description: as for outcome 2
Time Frame: Preoperative Visit (Day -30 to Day -1), Month 1, Month 3
Population: Consistent Cohort Analysis Set: All eyes in the FAS that have manifest refraction data at all post-operative visits from one month up to and including the visit where refractive stability is established.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 163
Number analyzed (eyes) | 326
percentage of eyes | 99.4

5. Primary Outcome: Percentage of Eyes With BCDVA Worse Than 20/40 (With BCDVA 20/20 or Better Preoperatively) at Refractive Stability
Description: VA was assessed using ETDRS charts at a distance of 4 meters with correction in place. BCDVA was measured in Snellen, where 20/20 indicates normal distance eyesight. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive stability was considered to be achieved at the Month 3 visit. A lower percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Day -30 to -1 (preoperative), up to Month 3
Population: SAS with requisite data at Month 3. Note: 1 eye was excluded from this analysis due to not having a preoperative BCDVA of 20/20 or better.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 165
Number analyzed (eyes) | 329
percentage of eyes | 0.0

6. Primary Outcome: Percentage of Eyes With BCDVA Loss of 2 Lines (10 Letters) or More From Preoperative Visit at Refractive Stability
Description: VA was assessed using ETDRS charts at a distance of 4 meters with correction in place and measured in logarithm Minimum Angle of Resolution, where each line on the letter chart represents 0.1 Snellen and 0.0 logMAR equates to 20/20 Snellen, or normal distance eyesight. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive stability was considered to be achieved at the Month 3 visit. A lower percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Day -30 to -1 (preoperative), up to Month 3
Population: SAS with requisite data at Month 3
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 165
Number analyzed (eyes) | 330
percentage of eyes | 0

7. Primary Outcome: Percentage of Eyes With Increase of Manifest Refractive Astigmatism Greater Than 2.00 Diopter (D) of Absolute Cylinder Compared to Preoperative Visit at Refractive Stability
Description: Manifest refractive astigmatism is the cylindrical portion of the subjective refraction. It is measured with ETDRS charts at a distance of 4 meters. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive stability was considered to be achieved at the Month 3 visit. A lower percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Day -30 to -1 (preoperative), up to Month 3
Population: SAS with requisite data at Month 3
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 165
Number analyzed (eyes) | 330
percentage of eyes | 0.0

8. Primary Outcome: Percentage of Eyes With Non-flap Related Ocular Serious Adverse Events at Refractive Stability
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test product). Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at Month 3 after surgery when compared with the Month 1 visit) that meets all the protocol-specified stability requirements. Refractive stability was considered to be achieved at the Month 3 visit. A lower percentage indicates a better outcome. Both eyes contributed data to this analysis. No hypothesis testing was pre-specified for this endpoint. This is a co-primary endpoint.
Time Frame: Up to Month 3
Population: SAS with requisite data at Month 3
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 165
Number analyzed (eyes) | 330
percentage of eyes | 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to approximately 1 year.
Description: AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting group.
Groups:
- Pretreatment: AEs in this group occurred prior to treatment with the WaveLight EX500 excimer laser with InnovEyes software in conjunction with InnovEyes sightmap
- WaveLight EX500 Excimer Laser System (Ocular): AEs in this group occurred after attempted treatment with the WaveLight EX500 excimer laser with InnovEyes software in conjunction with InnovEyes sightmap and include ocular events in the study eye
- WaveLight EX500 Excimer Laser System (Systemic): AEs in this group occurred after attempted treatment with the WaveLight EX500 excimer laser with InnovEyes software in conjunction with InnovEyes sightmap and include overall systemic events
Arm/Group | Pretreatment | WaveLight EX500 Excimer Laser System (Ocular) | WaveLight EX500 Excimer Laser System (Systemic)
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/336 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/168 | 4/336 | 0/168
Other Adverse Events (participants affected / at risk) | 3/168 | 0/336 | 10/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=168) | WaveLight EX500 Excimer Laser System (Ocular) (N=336) | WaveLight EX500 Excimer Laser System (Systemic) (N=168)
Retinal Tear (Eye disorders) | 0 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 2 | 0
Corneal opacity (Eye disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=168) | WaveLight EX500 Excimer Laser System (Ocular) (N=336) | WaveLight EX500 Excimer Laser System (Systemic) (N=168)
Corona virus infection (Infections and infestations) | 3 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to study.

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT04219891/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04219891/SAP_001.pdf